CLINICAL TRIAL: NCT06878872
Title: Adapting an Adolescent Weight Management Program for a Type 1 Diabetes Population
Brief Title: Type 1 Diabetes Adolescents for Healthier Lifestyles Study
Acronym: T1DAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K23DK132457 (NIH); 5K23DK132457 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes; Eating Behavior; Adolescent Obesity
Keywords: Teenagers; Diabetes; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Feeding Behavior; Pediatric Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1DAL Program (Experimental): Adolescent intensive health behavior and lifestyle treatment adapted for a type 1 diabetes population
  Interventions: Behavioral: T1DAL Program
- Usual Care (No Intervention): Adolescents continue their typical diabetes treatment management.

INTERVENTIONS:
Behavioral: T1DAL Program — T1DAL is a 16-week behavioral program. Teens meet in virtual groups and individually with a health coach throughout the program. Teens learn healthy lifestyle behaviors specific to living with type 1 diabetes and get opportunities to connect with other teens who are living with type 1 diabetes.
  Arms: T1DAL Program

SUMMARY:
Before the 1990s, obesity was rare among young people with type 1 diabetes (T1D), but now it is more common. Recent studies show that over 50% of young people with T1D will have overweight or obesity within five years of being diagnosed with T1D. Both obesity and T1D increase the risk of heart disease, and combined, these risks are even higher. Intensive health behavior and lifestyle treatments (IHBLTs) are proven to be effective for treating childhood obesity. However, managing T1D creates unique challenges that require adjustments to these treatments. For example, people with T1D need to eat even when they're not hungry to treat low blood sugar, blood sugar changes can make exercise harder, and some recommended "free foods" are high in unhealthy fats. Young people with T1D are also more likely to develop eating disorders. There is a need for IHBLTs that address these specific challenges and focus on preventing eating disorders in this group.

To address these needs, we developed the Type 1 Diabetes Adolescents for healthier Lifestyles (T1DAL) program, based on feedback from teenagers with T1D, their parents/caregivers, and pediatric endocrinologists. The goal of this study is to test whether the T1DAL program can improve the health and wellbeing of teens compared to usual care.

In this study, about 50 teens will be randomly assigned to either the T1DAL program or to Usual Care. Those in the T1DAL group will take part in a 16-week program designed specifically for teens with T1D to improve eating habits and diabetes management. Those in the Usual Care group will continue with their regular endocrinology appointments. At the end of the study, the Usual Care group will be offered a shortened version of the T1DAL program. All participants will have their height, weight, blood glucose, eating habits, diabetes management behaviors, and mood measured at the start and end of the study. They will also answer questions to track unhealthy eating and weight control behaviors over time. Additional analyses will look at factors that may lead to these behaviors in real life.

This project builds on Dr. Warnick's previous work in pediatric obesity and T1D, and it supports the NIDDK's goal of reducing diabetes-related heart problems. T1DAL could become an important public health program to improve the health of teens with T1D.

DETAILED DESCRIPTION:
Obesity was rare in youth with type 1 diabetes (T1D) prior to the 1990s, but the prevalence now exceeds that of youth in the general population. Recent studies indicate that over 50% of youth with T1D will develop overweight/obesity within five years of diagnosis. Obesity and T1D are individually associated with risks for cardiovascular disease, and combined, those risks are amplified. Intensive health behavior and lifestyle treatments (IHBLTs) are evidence-based, first-line treatments for pediatric obesity. Yet, there are unique challenges associated with managing T1D that require thoughtful adaptations to these IHBLTs. Challenges include needing to eat regardless of hunger to treat hypoglycemia, blood glucose changes making physical activity difficult, and recommended "free foods" that are high in saturated fats. Adolescents with T1D are also at high risk of developing disordered eating behaviors. There is a critical need for IHBLTs that address barriers specific to T1D and incorporate attention to eating disorder prevention in this at-risk population. Based upon multiple rounds of qualitative feedback from adolescents with T1D, their caregivers, and pediatric endocrinologists, our team developed the Type 1 Diabetes Adolescents for healthier Lifestyles (T1DAL) Study. The objective of this study is to test whether the T1DAL program preliminarily improves adolescents' health and wellbeing compared to a usual care control group.

In this study, approximately 50 total adolescents will be randomly assigned either to the T1DAL program or to Usual Care. Adolescents randomized to the T1DAL program will complete a 16-week IHBLT adapted to a T1D population. Those randomized to Usual Care will attend their routine endocrinology appointments. At the end of the study, those assigned to Usual Care will be offered an abbreviated T1DAL program. All adolescents' height, weight, time in target blood glucose range (70-180mg/dL), eating behaviors, diabetes management behaviors, and mood will be assessed at the start and end of study involvement. Participants will also complete ecological momentary assessments (EMA) at the start and end of study involvement to determine potential events of maladaptive eating and weight control behaviors over time. Exploratory analyses will evaluate correlates of these maladaptive eating and weight control behaviors in real-world settings.

This project builds upon Dr. Warnick's prior work in pediatric obesity and T1D. The proposed project aligns with the NIDDK's mission to mitigate diabetes-related cardiovascular events and has the potential to be an important public health intervention to improve the health of adolescents with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Teen diagnosed with type 1 diabetes at least 6 months ago
* Teen's body mass index greater than or equal to the 70th percentile for age and sex
* Teen lives with parent/caregiver
* Teen has access to a smart phone
* Teen and caregiver speak and write in fluent English

Exclusion Criteria:

* Teen has a medical condition that precludes them from participating in a group activity and/or any physical activity
* Teen experiencing psychosis or suicidality
* Teen lost a significant amount of weight in the 3 months prior to the study
* Teen currently in another intensive health behavior and lifestyle treatment and/or sees a dietician more than once per month on average
* Teen currently or planning to become pregnant
* Teen unwilling to wear a continuous glucose monitor for assessments
* Teen taking a medication known to impact weight and/or appetite

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
BMI Change | baseline, 4-months
  Change in body mass index
Time in Range Change | baseline, 4-months
  Change in time in the recommended glucose range (70-180 mg/dL)

SECONDARY OUTCOMES:
Events of Unhealthy Weight Control Behaviors | baseline, 4-months
  Events of maladaptive/disordered weight-control behaviors

OTHER OUTCOMES:
Correlates of Unhealthy Weight Control Behaviors | baseline, 4-months
  Environment cues, social cues, and affect via EMA survey

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Warnick, PhD, Principal Investigator — The Miriam Hospital

IPD SHARING:
Plan to Share IPD: No
Please contact the PI for a request of de-identified data.

DOCUMENTS (1):
  • Informed Consent Form (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT06878872/ICF_000.pdf